CLINICAL TRIAL: NCT03659734
Title: Randomized Controlled Trial to Evaluate the Relative Efficacy of Motivational Interviewing and Guided Opioid Tapering Support vs. Enhanced Usual Care to Promote Opioid Cessation After Orthopedic Surgery
Brief Title: Motivational Interviewing and Guided Opioid Tapering Support to Promote Postoperative Opioid Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jennifer Hah, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-43163; 1R01DA045027-01A1 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-09-06 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Opioid Cessation
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing and Guided Opioid Tapering Support (Experimental)
  Interventions: Behavioral: Motivational Interviewing and Guided Opioid Tapering Support
- Enhanced Usual Care (Experimental)
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Motivational Interviewing and Guided Opioid Tapering Support — Following surgery, participants will undergo motivational interviewing with a trained member of the study staff. These calls will occur weekly for 6 weeks with a follow-up call at 10 weeks or until the participant completes the protocol.
  Arms: Motivational Interviewing and Guided Opioid Tapering Support
Behavioral: Enhanced Usual Care — Following surgery, participants will receive phone calls from a trained member of the study staff to discuss various aspects of surgical recovery and medication use. These calls will occur weekly for 6 weeks with a follow-up call at 10 weeks or until the participant completes the protocol.
  Arms: Enhanced Usual Care

SUMMARY:
The purpose of this study is to evaluate the relative efficacy of enhanced usual care versus motivational interviewing and guided opioid tapering support to promote opioid cessation after total hip or knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planning to undergo surgery
* English speaking
* Ability and willingness to complete questionnaires and assessments
* Scheduled for total hip, knee, or shoulder replacement
* Preoperative opioid use and opioid use 14 days after surgery to increase the likelihood of delayed opioid cessation.
* Not under the care of a current pain management provider

Exclusion Criteria:

* Any conditions causing inability to complete assessments
* Known pregnancy
* Elevated suicidality
* Enrollment in conflicting perioperative trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2024-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hah, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Interviewing and Guided Opioid Tapering Support | Enhanced Usual Care
Started | 87 | 92
Completed | 87 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing and Guided Opioid Tapering Support | Enhanced Usual Care | Total
Number analyzed (Participants) | 87 | 92 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (14.0) | 57.2 (23.2) | 59.4 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 64 | 119
  Male | 32 | 28 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 79 | 86 | 165
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 4 | 9
  White | 68 | 76 | 144
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 2 | 3 | 5
Numeric Rating Scale of Pain [Mean (Standard Deviation); unit: units on a scale] — Total range from 0 to 10 with 0 being no pain and 10 being the worst pain imaginable.
  units on a scale | 3.3 (2.9) | 2.8 (2.8) | 3.0 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Time to Opioid Cessation
Description: Time to opioid cessation between the two groups will be analyzed using survival analysis
Time Frame: Through study completion, an average of 1 year
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Motivational Interviewing and Guided Opioid Tapering Support | Enhanced Usual Care
Number analyzed (Participants) | 87 | 92
days | 28 [14 to 49] | 25 [15 to 51]

2. Secondary Outcome: Number of Participants With Opioid Misuse (Postoperative COMM Score Greater Than or Equal to 9)
Description: Assessed by total score on the Current Opioid Misuse Measure (COMM). The Current Opioid Misuse Measure is a self-report measure of risk for aberrant medication related behavior among persons who are prescribed opioids for pain. The COMM contains 17 items rated from 0="never" to 4="very often" . The 17 items are summed to create a total score with a minimum of 0 to a maximum of 68. Higher scores represent a higher risk of potential opioid medication misuse (worse outcome). Patients exhibiting opioid misuse (binary outcome) were defined as those reporting a postoperative COMM score greater than or equal to 9.
Time Frame: Through study completion, 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing and Guided Opioid Tapering Support | Enhanced Usual Care
Number analyzed (Participants) | 87 | 92
Participants | 20 | 17

ADVERSE EVENTS:
Time Frame: For 1 year after surgery
Arm/Group | Motivational Interviewing and Guided Opioid Tapering Support | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/92
Other Adverse Events (participants affected / at risk) | 0/87 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT03659734/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03659734/SAP_001.pdf
  • Informed Consent Form (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03659734/ICF_002.pdf